CLINICAL TRIAL: NCT00727090
Title: Use of Conivaptan (Vaprisol) for Hyponatremic Neuro-ICU Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment below goal.
Sponsor: Northwestern University (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Andrew Naidech, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1507-10
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2010-09-27 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Hyponatremia
MeSH Terms: conditions — Hyponatremia | interventions — conivaptan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Conivaptan in addition to usual care at the discretion of the attending medical staff
  Interventions: Drug: Conivaptan
- 2 (No Intervention): Usual care by the attending physician staff

INTERVENTIONS:
Drug: Conivaptan — Conivaptan 20 mg once, followed by conivaptan 20 mg over 24 hours
  Other Names: Vaprisol
  Arms: 1

SUMMARY:
Conivaptan (Vaprisol) is FDA-Approved for the treatment of low serum sodium (hyponatremia), but there are few data in patients with neurologic disease. Very low serum sodium in patients with brain injury can be life-threatening and is associated with cerebral edema (swelling of brain tissue). This can be important in patients with brain hemorrhage, brain tumors, or stroke (cerebral infarction).

This is a pilot study to test the hypothesis that conivaptan (Vaprisol) leads to a greater increase in sodium than usual care. Patients will be randomly assigned to usual care or the lower FDA-approved dose of conivaptan (Vaprisol). We will track the use of other interventions, such as the use of hypertonic saline (concentrated salt solution), diuretics and salt tablets. A blinded co-investigator will record neurologic examination results (NIH Stroke Scale and Glasgow Coma Scale).

ELIGIBILITY:
Inclusion Criteria:

* severe hyponatremia (Na < 130 mmol/L) or
* symptomatic hyponatremia - Na < 135 mmol/L for at least six hours with Glasgow Coma Scale < 15

Exclusion Criteria:

* Enrollment in the NMH high-risk spine protocol. These patients receive large amounts of fluids, have rapid changes in electrolytes, and are typically corrected in 48 hours
* Expected death from any cause
* Known sensitivity or allergy to conivaptan
* Renal failure (baseline creatinine > 1.5 mg/dL)
* Clinical diagnosis of hypovolemia, or by central venous pressure (CVP) < 5 mm Hg if a central venous catheter is in place
* Concomitant use of potent inhibitors of cytochrome P-450 isoenzyme 3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir). These agents are not commonly used in the Neuro-ICU
* Clinical diagnosis of liver failure or insufficiency
* Pregnancy (must be excluded before entry)
* Lack of informed consent from the patient or a legally authorized representative (LAR)
* Use of intra-arterial vasodilators (e.g. verapamil, nicardipine) within 24 hours (e.g. for vasospasm after SAH)
* Concern by the Neuro-ICU pharmacist of a drug-drug interaction that would meaningfully impact care (the Neuro-ICU pharmacist will review the medication regimen before recruitment)
* Patients with a diagnosis of diabetes insipidus or treated with vasopressin, since these patients are already treated for abnormal free water balance
* Patients with congestive heart failure, since this is an approved use of the drug (these patients are typically not cared for in the Neuro-ICU)
* Age<18 years (these patients are not cared for at NMH)
* Inclusion declined by the attending physician or consulting study nephrologist

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Naidech, MD, MSPH, Principal Investigator — Northwestern University

REFERENCES:
- [Derived] Naidech AM, Paparello J, Liebling SM, Bassin SL, Levasseur K, Alberts MJ, Bernstein RA, Muro K. Use of Conivaptan (Vaprisol) for hyponatremic neuro-ICU patients. Neurocrit Care. 2010 Aug;13(1):57-61. doi: 10.1007/s12028-010-9379-5. PMID 20568023

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Conivaptan: Conivaptan per package labeling, 20 mg IV bolus followed by 20 mg IV infusion over 24 hours
- Usual Medical Care: Usual care by the attending physician staff
Period: Overall Study
Arm/Group | Treatment: Conivaptan | Usual Medical Care
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment: Conivaptan | Usual Medical Care | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (22.0) | 67 (2) | 55 (19.2)
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 70 years | 3 | 3 | 6
  >70 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Sodium From Baseline to 6 Hours
Time Frame: 48 hours
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: mMol/L
Arm/Group | Treatment: Conivaptan | Usual Medical Care
Number analyzed (Participants) | 3 | 3
mMol/L | 7 (1.7) | -0.6 (2.1)
Statistical Analysis 1: Comparison: Treatment: Conivaptan; Null Hypothesis: Change in serum sodium from baseline is not different between groups; Test type: Non-Inferiority or Equivalence — Equivalence; p < 0.05, t-test, 2 sided

2. Secondary Outcome: NIH Stroke Scale
Description: Standardized neurologic examination, ranging from 0 (best) to 42 (worst possible).
Time Frame: 48 hours
Population: Comparison of distribution; n enrolled was insufficient and trial was halted for poor recruitment.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Conivaptan: Conivaptan in addition to usual care at the discretion of the attending medical staff
  Conivaptan: Conivaptan 20 mg once, followed by conivaptan 20 mg over 24 hours
- Usual Care: Usual care by the attending physician staff
Arm/Group | Conivaptan | Usual Care
Number analyzed (Participants) | 3 | 3
score on a scale | 19 [17 to 21] | 12 [8 to 14]

3. Secondary Outcome: Glasgow Coma Scale
Description: Standardized examination of mental status ranging from 3 (worst) to 15 (best possible)
Time Frame: 48 hours
Population: all enrolled patients
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Conivaptan | Usual Care
Number analyzed (Participants) | 3 | 3
score on a scale | 9 [9 to 10] | 12 [12 to 13]

4. Other Pre Specified Outcome: Change in Serum Sodium From Baseline to 12 Hours
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: mMol/L
Arm/Group | Treatment: Conivaptan | Usual Medical Care
Number analyzed (Participants) | 3 | 3
mMol/L | 7.7 (4.0) | 1.7 (0.6)

5. Other Pre Specified Outcome: Change in Serum Sodium From Baseline to 18 Hours
Time Frame: 18 hours
Measure: Mean (Standard Deviation); unit: mMol/L
Arm/Group | Treatment: Conivaptan | Usual Medical Care
Number analyzed (Participants) | 3 | 3
mMol/L | 7.3 (4.0) | 1.3 (2.1)

6. Other Pre Specified Outcome: Change in Serum Sodium From Baseline to 24 Hours
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mMol/L
Arm/Group | Treatment: Conivaptan | Usual Medical Care
Number analyzed (Participants) | 3 | 3
mMol/L | 9.7 (3.2) | 0 (1)

7. Other Pre Specified Outcome: Change in Serum Sodium From Baseline to 36 Hours
Time Frame: 36 hours
Measure: Mean (Standard Deviation); unit: mMol/L
Arm/Group | Treatment: Conivaptan | Usual Medical Care
Number analyzed (Participants) | 3 | 3
mMol/L | 8 (5.6) | -1.7 (2.1)

8. Other Pre Specified Outcome: Change in Serum Sodium From Baseline to 48 Hours
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mMol/L
Arm/Group | Treatment: Conivaptan | Usual Medical Care
Number analyzed (Participants) | 3 | 3
mMol/L | 6 (5) | -0.7 (3.2)

ADVERSE EVENTS:
Time Frame: 48 hours after study start
Description: Hypovolemia, clincial diagnosis by intensivist or central venous pressure < 5 mmg Hg; Hypotension, systolic BP < 100 mm Hg or requiring new vasopressors; Rash at study drug infusion site; New core temperature at least 100.4F;
Arm/Group | Treatment: Conivaptan | Usual Medical Care
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Conivaptan (N=3) | Usual Medical Care (N=3)
Hypotension (Cardiac disorders) | 2 (2) | 1 (1)
Hypovolemia (Cardiac disorders) | 1 (1) | 0 (0)
Fever (Infections and infestations) | 0 (0) | 2 (2) — New core temperature at least 100.4F

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less